CLINICAL TRIAL: NCT01225744
Title: A Phase II Study Evaluating the Use of Concurrent Cetuximab, Irinotecan, Oxaliplatin and UFT in the First Line Treatment of Patients With Metastatic Colorectal Cancer
Brief Title: Erbitux Study of CPT11, Oxaliplatin, UFToral Targeted Therapy
Acronym: eSCOUT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Suzanne Rowland, Clinical Trials Project Manager, The Christie NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07_DOG03_133
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; Oxaliplatin; Tegafur; Uracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab plus Irinotecan, Oxaliplatin and UFT (Experimental): Cetuximab plus Irinotecan, Oxaliplatin, UFToral
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: UFT

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be prepared under Good Manufacturing practice (GMP) and supplied by Merck KGaA (Darmstadt, Germany) as a solution for intravenous infusion. It will be made up into 250ml with N/Saline.
  Dose administered is 400mg/m2 and will be given on day 1 and day 15 of a 28 day cycle.Cetuximab will always be administered first, i.e. the cetuximab infusion should be completed one hour before any chemotherapy begins. The cetuximab dose must always be based on the body surface area(BSA). There is no restriction for cetuximab in patients with a BSA > 2 m2 .
  Other Names: Erbitux
Drug: Irinotecan — Dose is 180mg/m2 made up into 250ml with 5% dextrose or 0.9% saline. It will be administered as a short infusion over 60-90 minutes after a 60 minute gap left after cetuximab administration. Irinotecan is administered on day 1 of the 28 day cycle.
  Other Names: Camptosar
Drug: Oxaliplatin — Dose is 100mg/m2 and will be made up into 250ml with 5% dextrose. It will be administered as a short infusion over 120 minutes after the 60 minute gap left after cetuximab administration. Oxaliplatin is administered on day 15 of the 28 day cycle.
  Other Names: Eloxatin
Drug: UFT — UFT dose is 250mg/m2 and is given in three divided doses with calcium folate 30mg p.o. tds on days 1-21 of the 28 day cycle. The highest dose of UFT should be given in the morning if the dose cannot be divided equally.
  Other Names: Tegafur; Uracil

SUMMARY:
A Phase II trial to demonstrate the response rate, using the Response evaluation criteria in solid tumours (RECIST) criteria, of patients with locally advanced / metastatic colorectal cancer treated with combination of irinotecan, oxaliplatin, UFT and cetuximab.

ENDPOINTS Primary: Objective response rate (RECIST) Secondary: Progression free survival (PFS), Overall survival (OS) Toxicity (CTCAE), Resectability of liver, lung and pelvic disease after chemotherapy, Time to progression (TTP).

POPULATION: The trial aims to recruit 50 patients with inoperable, metastatic colorectal cancer ELIGIBILITY: Histologically confirmed colorectal adenocarcinoma Normal haematology and adequate renal and liver function Written informed consent and able to attend follow-up for at least 3 months TREATMENT 4 weekly cycles of chemotherapy with alternating irinotecan (day 1) and oxaliplatin(day 15). Cetuximab every 2 weeks and oral UFT with Leucovorin for 3 weeks every 4 weeks.

DURATION First patient recruited April 2009. Accrual to take place over 24 months Follow-up will continue until death or for a minimum of 3 years

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum.
* Patients must not have a mutation of K-ras
* Inoperable metastatic or locoregional disease (synchronous or recurrence)
* No previous chemotherapy for established metastatic disease (adjuvant chemotherapy must have been completed more than 6 months prior to trial entry)
* Measurable or evaluable disease
* Bone marrow function: neutrophil count >1.5 x109/l and platelet count >150 x109/l
* Hepatobiliary function: serum bilirubin <1.5 x upper limit of normal (ULN); ALP <5 x ULN; transaminase (AST or ALT) <3 x ULN.(≤ 5 if liver mets are present)
* Renal function: estimated creatinine clearance >50 ml/min, or measured Glomerular filtration rate (GFR) (EDTA or creatinine clearance) in normal range
* ECOG performance status 0-1 and considered fit and able to undergo all possible treatments
* For women of child-bearing potential a negative pregnancy test is required and adequate contraceptive precautions such as a sheath for their partner must be used
* For men - adequate contraception such as a sheath must be used
* Patients must give written, informed consent
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Patients that have a K-ras mutation
* Concurrent uncontrolled medical illness, or other previous or current malignant disease likely to interfere with protocol treatments or comparisons
* Partial or complete bowel obstruction
* Prior EGFR antibody therapy
* Age <18
* Chronic diarrhoea or inflammatory bowel disease
* Known Pyruvate Dehydrogenase Phosphatase (DPD) deficiency
* Gilbert's syndrome or other congenital abnormality of biliary transport
* Previous transplant surgery, requiring immunosuppressive therapy
* Regular / uncontrolled angina or cardiac arrhythmias
* Clinically relevant coronary artery disease. History of Myocardial infarction in the last 12 months
* Previous investigational agent in the last 4 weeks
* Metastatic disease to brain
* Any pregnant or lactating women
* Patients receiving therapy with haloginated antiviral drugs (eg: sorivudine)
* Patients who have experienced life-threatening toxicities with fluoropyrimidines treatment
* Patients suffering from any condition that may affect the absorption of UFT or folinic acid.
* Patients with known deficiency of or are on inhibitors of cytochrome P450 2A6
* Patients who have previously had radiotherapy to the abdomen or pelvis in the last 6 months
* Any medical or psychological condition that in the opinion of the investigator would not enable the patient to complete the study or knowingly give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Objective response rate (according to RECIST criteria) | 8 weeks post starting treatment
  Patients will receive triphasic CT scans at 8 weekly intervals after treatment has started. Patients remain on trial until disease progression or at the discretion of the Investigator.

SECONDARY OUTCOMES:
Progression Free Survival | 8 week intervals post starting treatment
  Progression will be defined according to RECIST criteria with appropriate clinical assessment and radiological investigations. This will be measured from the time of entry into the study.
Overall survival (OS; all causes of death). | 3 years post treatment
  The date and cause of death will be recorded for each patient. Survival will be measured from the date of registration into the trial and will be reported on an intention-to treat-basis.
Toxicity | 2 months post starting treatment
  Grade 3 or 4 Adverse Events experienced from the start of treatment up to the point of the first response CT scheduled for 8 weeks after treatment start date.
  Number and description of Serious Adverse Events experienced will also be recorded.
Resectability of liver, lung and pelvic disease after chemotherapy | 8 weekly intervals from the start of treatment
Time to progression (TTP) | 8 weekly intervals following starting treatment
  This is defined as the time from start of treatment to the time of documented radiological progression of disease locally

CONTACTS AND LOCATIONS:
Overall Officials: Mark Saunders, Principal Investigator — Christie NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - North Wales Cancer Treatment Centre, Llansantffraid Glan Conwy
  - The Royal Marsden, London and Surrey
  - The Christie NHS Foundation Trust, Manchester